CLINICAL TRIAL: NCT05013606
Title: Hydrogen Water as a Treatment for Chronic Fatigue Syndrome: A Pilot Study
Brief Title: Hydrogen Water Treatment for Chronic Fatigue Syndrome
Acronym: H2CFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Fred Friedberg, Research Associate Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H2CFSPilot 1241294
Record Dates: First submitted 2019-02-27; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Chronic Fatigue Syndrome
Keywords: hydrogen; treatment
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Water

STUDY DESIGN:
Intervention Model Description: This clinical study involves two groups, one group receiving only the active treatment, hydrogen pills mixed with water, and the other group receiving only a placebo pill mixed with water.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Pills for both conditions look very similar and each group sees only the pill assigned to that group (H2 or placebo) and not the pill assigned to the other group. Also neither the outcome assessor nor the investigator know which condition that specific individual subjects are assigned to. This is because a blocked randomization schedule of numbers (1s and 2s) is used to assign each consecutive subject enrolled in the study to one of the study conditions. The code that links each subject to an identifiable condition assignment is known only by the PI and not the staff who selects the pills to be sent out to each subject or by the outcomes assessor. Also the subject fills out online outcome forms that involve no interaction with study staff, thus avoiding any staff-specific influence on online outcome forms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment: Hydrogen water (Experimental): Hydrogen pills mixed in a water glass that is ingested up to five time a day for 30 days.
  Interventions: Dietary Supplement: Hydrogen water
- Placebo: Inactive pill (Placebo Comparator): Inactive pills mixed in a water glass that is ingested up to five time a day for 30 days.
  Interventions: Dietary Supplement: Hydrogen water

INTERVENTIONS:
Dietary Supplement: Hydrogen water — This is an over the counter pill supplement that is dissolved in water.

SUMMARY:
The proposed placebo-controlled pilot study will examine hydrogen water as a treatment for myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS). 25 subjects who meet strict criteria for ME/CFS will be recruited. The 30 day trial will involve subjects ingesting 1-5 8 oz. glasses of hydrogen-dissolved water per day. The placebo condition will involve the same daily ingestion schedule but with an inert placebo pill instead of the active hydrogen treatment pill. The proposed study is intended to establish feasibility of the clinical protocol and examine potential treatment effects of hydrogen water which may include symptom reduction and possibly improved functioning. If feasibility and apparent treatment effects are confirmed, a large clinical trial will be proposed for submission to NIH. In addition to potential therapeutic properties, H2 water is portable, easily administered and safe to ingest.

Self-report assessments for ME/CFS symptoms, fatigue, autonomic symptoms, physical function, anxiety, and depression will be done in the week before and the week after the 30 day trial. In addition, 7-day home-based objective assessments of heart rate variability (a measure of parasympathetic function) and accelerometry (a physical activity assessment) will be scheduled before and after the intervention period.

DETAILED DESCRIPTION:
SPECIFIC AIMS

The aim of this pilot randomized control trial (RCT) is to explore the possible beneficial effect of a novel therapy, molecular hydrogen (H2) for the symptoms and related functional limitations in patients with chronic fatigue syndrome.

BACKGROUND AND SIGNIFICANCE Oxidative stress and impaired energy metabolism have been implicated in the pathophysiology of myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS), a debilitating illness without clearly identified etiology or effective medical treatments. As such, treatments that reduce oxidative stress and yield improvements in energy production may show potential to ameliorate the symptoms and functional limitations of this illness. Numerous publications on the biological and medical benefits of H2 have shown that H2 reduces oxidative stress not only by direct reactions with strong oxidants, but also indirectly by regulating various gene expressions. In addition to its potential therapeutic properties for ME/CFS, H2 water is portable, easily administered and safe to ingest.

PRELIMINARY STUDIES

The proposed study is a pilot study in ME/CFS for which there are no directly applicable preliminary studies utilizing the proposed H2 therapy.

RESEARCH DESIGN AND METHODS

Eligible subjects will be recruited by advertising. Assessments will be conducted by telephone, via home-based monitoring, and online diaries. The PI has 16 years' experience recruiting ME/CFS patients for his NIH funded studies. Given the absence of effective interventions for this illness and the absence of in-person visits in the proposed study, the possibility of being helped by the benign treatment of H2 is likely to attract many patients with ME/CFS.

Study Sample

Subjects who meet the inclusion/exclusion criteria below and provide consent will be recruited and randomized sequentially 1:1 to receive either H2 or placebo. The investigators will seek to enroll a total of 25 patients meeting enrollment criteria and randomized to H2 vs placebo arms. The investigators project a study duration of 8-10 months.

Screening

Inclusion criteria: These are: patients aged 18-65 of both sexes considered physically capable and willing to perform the study tasks, including wearing a heart monitor and an actigraph (at baseline and post-treatment weeks). Subjects must also meet our validated phone-screen eligibility for ME/ CFS criteria. A physician note confirming a CFS diagnosis will be requested.

Medical exclusions, determined by validated phone screen interview, will consist of cases of fatigue clearly attributable to self-report medical conditions such as untreated hypothyroidism, unstable diabetes mellitus, organ failure, chronic infections, and chronic inflammatory diseases, or AIDS. Exclusionary psychiatric disorders include any psychosis, or alcohol/ substance abuse within two years prior to illness onset and any time afterward, and current or past depression with melancholic or psychotic features within 5 years prior to onset of ME/CFS or anytime afterward. Pregnancy, as determined by reliable home test kit sent to subjects, is also an exclusion. Two other exclusionary criteria will be used: a) patients on heart medication or patients not dose-stabilized for at least 3 months on antidepressant drugs; b) patients at significant risk of suicide or in need of urgent psychiatric treatment. As much as possible, appropriate medical and psychiatric referrals to facilities local to subjects will be provided.

Procedures/Outcome measures

This will be a double blinded, placebo-controlled trial. Subjects will be sequentially randomized in a 1:1 ratio to receive H2, or corresponding placebo, additional to all standard-of-care treatments. All study-related participant activities, including questionnaires, activity and heart monitoring, and online diaries will be completed by participants in their homes. No face-to-face visits to Stony Brook are involved. H2 water is Generally Recognized As Safe (GRAS) and is increasingly available on the general consumer market. Self-report questionnaire assessments for ME/CFS symptoms, fatigue, autonomic symptoms, physical function, anxiety, and depression will be done in the week before and the week after the 30 day trial. In addition, an online web diary to record ME/CFS symptoms and home-based objective assessments of heart rate variability (a measure of parasympathetic function) and accelerometry (a physical activity assessment) will be scheduled before, during, and/or after the intervention period.

STATISTICS The study will define improvement by a 50% reduction in ME/CFS symptoms. Repeated measures analysis of variance (ANOVA) will compare pre- and post-treatment measurements of effectiveness and general health markers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic fatigue, chronic fatigue syndrome, ME/CFS or something similar.
* age 21-65

Exclusion Criteria:

* Other major medical condition or regular medication that produces fatigue.
* No home computer
* No internet access

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 4 weeks
  Fatigue Severity Scale; Minimum value=1; Maximum value=7; Range: 1.00-7.00. Higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | 4 weeks
  Self-report measure of sleep quality; A patient's seven subscores, each of which can range from 0 to 3 are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Short Form-36 Physical Function Subscale | 4 weeks
  Self-report measure of physical functioning. The Short Form 36 physical function subscale is composed of ten items encompassing a hierarchical range of difficulties. Each item is scored on the basis of the limitations perceived by surveyed individuals. Item scores (1, 2, or 3) are summed to obtain a total score, which can then be scaled relative to its range. Higher scores indicate higher physical function.
Depression, Anxiety, and Stress Scale | 4 weeks
  Self-report measure of depression, anxiety and stress symptoms; This 21-item stress measure contains three seven-item subscales: anxiety, depression and stress. Domain scores are calculated by summing all items in a domain and multiplying by two.
  Scores range from 0-37+ on each subscale with higher scores indicated greater symptom severity.

OTHER OUTCOMES:
Heart rate variability | 7 weeks
  Objective measure of autonomic function
Salivary C-Reactive Protein | 6 weeks
  This commonly used objective marker of systemic inflammation can be assessed in salivary samples.
Salivary Uric Acid | 6 weeks
  Salivary uric acid is a measure of antioxidant status.
Salivary Alpha Amylase | 6 weeks
  This digestive enzyme appears to be a reliable marker of sympathetic nervous activity

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University, Stony Brook, New York, United States